CLINICAL TRIAL: NCT01054066
Title: Management of Chronic Kidney Disease in Eastern North Carolina (MARKER)
Brief Title: Managing Chronic Kidney Disease in Eastern North Carolina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: The Kate B. Reynolds Charitable Trust (Other)
Responsible Party: Principal Investigator, Paul Bolin, Chair of Internal Medicine, East Carolina University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008-317
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Cardiovascular Disease; Hypertension; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Hypertension; Anemia | interventions — Primary Health Care; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Chronic Kidney Disease Education — Instituting teaching programs to manage hypertension, diabetes, anemia, proteinuria and cardiovascular disease in patients.
  Other Names: primary care; primary care clinics; education

SUMMARY:
The purpose of this program is to educate primary care physicians in four underserved clinics in eastern North Carolina about chronic kidney disease.

DETAILED DESCRIPTION:
The Division of Nephrology within the Brody School of Medicine recently form a center to focus attention on the needs of patients with kidney disease in eastern North Carolina. It is estimated that more than 40 million Americans have or at risk for CKD. The estimate for CKD in eastern North Carolina is exacerbated by poor access to health care. The mission of the East Carolina University Center for the Study and Treatment of Kidney Disease (ECCKD) is to increase education and awareness, improve treatment and outcomes through research, and better serve patients with CKD in eastern North Carolina.

ELIGIBILITY:
Inclusion Criteria:

* Primary care clinics in eastern North Carolina with a high penetration of chronic kidney disease, risk factors for chronic kidney disease and poverty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2008-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the effect of CKD education on the behavior of the primary care physician in underserved areas in Eastern North Carolina. | every 6 months

SECONDARY OUTCOMES:
To assess the rate of reduction of CKD in patients in Eastern North Carolina. | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bolin, MD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States